CLINICAL TRIAL: NCT03493581
Title: Precision Immuno-Oncology for Advanced Non-small Cell Lung Cancer Patients With PD-1 ICI Resistance (PIONeeR-BioMarkers (BM) Profiling)
Acronym: PIONeeR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2017-67; 2018-A03518-45 (Other: IDRCB)
Record Dates: First submitted 2018-03-20; First posted 2018-04-10 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Non-small Cell Lung Cancer Patients
MeSH Terms: interventions — Biopsy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NSCLC patients (Experimental)
  Interventions: Procedure: BIOPSY; Diagnostic Test: blood-sampled; Other: feces samples

INTERVENTIONS:
Procedure: BIOPSY — re-biopsy (primitive tumor or metastasis) specifically for the study, at V2(6 weeks)
Diagnostic Test: blood-sampled — * after 3 or 4 weeks (V1-1st assessment of PK/PD, after the 2d course),
  * after 6 weeks (V2),
  * after 8 or 9 weeks (V3-2nd assessment of PK/PD, after the last course),
  * - after 12 weeks of treatment (V4- samples for 3rd assessment of PK/PD and other analyses ).
  * after 18 weeks (V5- samples for 4th assessment of PK/PD and other analyses,),
  * after 24 weeks of treatment (V6-5th assessment of PK/PD and other analyses).
Other: feces samples — If they are amenable to collect feces samples at home, an auto collection kit will be supplied to them, before the first injection (Vs) and when they come for the 2nd course (i.e after 3 or 4 weeks post initiation) in order to self-collect feces within the week beforeV2 - 6 weeks post initiation).

SUMMARY:
PIONeeR study is a prospective, multicenter study without administration of an investigational product.

The promotion and funding will be done by the Assistance Publique Hôpitaux de Marseille (APHM), the coordination by AMU. There will be 3 principal investigational clinical centres in France:

* Service d'Oncologie Multidisciplinaire et Innovations Thérapeutiques in APHM, Marseille, supervised by Prof. L. Greillier
* Medical Oncology Department of Centre Léon Bérard, Lyon, supervised by Prof. M. Pérol
* Unité d'Oncologie Thoracique, CHU Larrey /Oncopôle, Toulouse, supervised by Prof. J. Mazières.

Some secondary centres, nearby the three principal mentioned above, will be associated to ensure recruitment of patients, in accordance to provisional planning.

* The primary objective is to validate the existence and distribution of the hypothetical immune profile (within blood and tumoral tissue) explaining primary or adaptive resistance to standard PD-1 inhibitors monotherapy, in NSCLC patients.
* The secondary objectives are to better characterize :

  * PK/PD relationships,
  * inter-patient PK variability,
  * If systemic exposure levels could be predictive of efficacy of PD-1 ICI, in NSCLC patients.
* Some exploratory objectives are :

  * to assess a predictive value of a panel of endothelial biomarkers, in NSCLC patients.
  * to compare predictive immune & endothelial biomarker profiles with those of sensitive tumors.
  * to better understand which profiles track significantly with progression following PD-1 ICI administration, in order to improve advanced NSCLC patients' stratification, for future clinical trials.

DETAILED DESCRIPTION:
Visits will match with usual schedule of patient's appointments with their referent oncologist or for injections of ICIs, when blood sampling or biopsies will be done. Feces will be collected by patients themselves, at home (optional).

The same day of registration for either an EMA approved first line PD-1 or PD-L1 inhibitor in combination with platinum-based chemotherapy OR a standard 2nd or 3rd line PD-(L) 1 ICIs monotherapy (to date, Nivolumab, Pembrolizumab, Atezolizumab), 450 advanced NSCLC patients will undergo a screening visit (Vs). If they are eligible, after signing an informed written consent, they will be blood-sampled specifically for the study:

* after 3 or 4 weeks (V1-1st assessment of PK/PD, after the 2d course),
* after 6 weeks (V2),
* after 8 or 9 weeks (V3-2nd assessment of PK/PD, after the last course),
* after 12 weeks of treatment (V4- samples for 3rd assessment of PK/PD and other analyses ).
* after 18 weeks (V5- samples for 4th assessment of PK/PD and other analyses,),
* after 24 weeks of treatment (V6-5th assessment of PK/PD and other analyses).

Patients will also be re-biopsied (primitive tumor or metastasis) specifically for the study, at V2. Referent patients'oncologist will opt for the simplest technical approach with a minimal risk exposure for patients. Standard procedures will be implemented for subsequent patient's monitoring.

Patients will also provide remaining samples from pre-treatment surgical resections/biopsies (primitive tumor or metastasis).

If they are amenable to collect feces samples at home, an auto collection kit will be supplied to them, before the first injection (Vs) and when they come for the 2nd course (i.e after 3 or 4 weeks post initiation) in order to self-collect feces within the week beforeV2 - 6 weeks post initiation).

Following the last study visit (V4 or V5 or V6)or at the time of a subsequent disease progression, patients will enter to the follow up period (a minimum 24 weeks ). They will be followed by their usual referent oncologist, no additional visit is required. Subsequent response to the anti-PD (L) 1 treatment, anti-cancer therapy, survival will be collected via patient medical records and analysed for current study.

ELIGIBILITY:
Inclusion Criteria:

* - Patients must be over 18 years
* Patients must have histologically confirmed diagnosis of advanced (proven stade IV) or recurrent NSCLC,
* Their ECOG Performance Status must be of 0 or 1
* EITHER patients must be previously untreated and eligible for an EMA approved first line PD-1 or PD-L1 inhibitor in combination with platinum-based chemotherapy, irrespective of their tumor histology
* These EMA approved first line combinations must be reimbursed by French Health Insurance or at least, must have an Authorization for Temporary Use (ATU) in France
* OR Patients must display disease progression after at least one line of platinum-based chemotherapy and eligible for a registered second or third line PD-1 or PD-L1 inhibitor in monotherapy (to date, Nivolumab, Pembrolizumab, Atezolizumab)
* For patients registered for a 2nd or 3rd line, those with known actionable molecular alteration (EGFR activating mutation, ALK rearrangement, ROS1 rearrangement) should have received a specific inhibitor
* Patients must have an available archived tissue from a standard tumor biopsy for PD-L1 assessment, done before PD-1 ICI initiation
* Patients must have an available archived tissue from a standard tumor biopsy for PD-L1 assessment, done before PD-1 ICI initiation
* Patients must have adequate organ functions
* Patients must have provided a signed and dated, written informed consent prior to any study specific procedures, sampling and analyses

Exclusion Criteria:

* Patients previously untreated and eligible for a first line PD-1 or PD-L1 inhibitor in monotherapy
* Combination of PD-1 or PD-L1 inhibitor with bevacizumab
* Exclusive bone progression
* Exclusive cerebral progression not amenable to surgical biopsy
* Absence of a target lesion according to RECIST criteria 1.1
* Life expectancy of less than 3 months
* Severe adverse events from PD-1 treatment
* Abnormal coagulation contraindicating biopsy
* History of hemorrhagic or thrombotic stroke, TIA or other CNS bleeds
* Active uncontrolled or serious infection (viral, bacterial or fungal)
* Active infection including VHB and VHC infections
* Individuals deprived of liberty or placed under the authority of a tutor
* Patient unable to understand, read and/or sign an informed consent
* Any condition which in the Investigator's opinion would jeopardize compliance with the protocol of the study
* Patients without Health insurance scheme or Universal Medical Coverage (CMU) or any equivalent scheme
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2018-03-08 (Actual); Primary Completion 2024-03-08 (Estimated); Study Completion 2024-08-12 (Estimated)

PRIMARY OUTCOMES:
Immuno-monitoring | 54 MONTHS
  BLOOD SAMPLES to characterize B, T, NK, and dendritic cell subsets and monocyte populations as well as Innate Lymphoid Cells (ILC) with cytometry analysis

SECONDARY OUTCOMES:
Measure the number of somatic mutations | 54 MONTHS
  BLOOD SAMPLES- extraction of nucleic acids from Plasma
Measure the number of somatic mutations | 54 MONTHS
  Tumor tissues- extraction of nucleic acids
measure the Circulating endothelial cells (CECs) | 54 MONTHS
  BLOOD SAMPLES using a CD146-based immunomagnetic separation assay.
Minimum Plasma Concentration Cmin of anti PD (L) 1 treatment | 54 MONTHS
  BLOOD SAMPLES
Maximum Plasma Concentration Cmax of anti PD (L) 1 treatment | 54 MONTHS
  BLOOD SAMPLES
lymphocytes DNA extraction's | 54 MONTHS
  Relevant polymorphisms will be screened by NGS technology

CONTACTS AND LOCATIONS:
Overall Officials: François CREMIEUX, Study Director — ASSISTANCE PUBLIQUE HOPITAUX D EMARSEILLE
Locations (1):
- Assistance Pubique Hopitaux de Marseille, Marseille, France